CLINICAL TRIAL: NCT03109041
Title: Initial Feasibility Study to Treat Resectable Pancreatic Cancer With the Permanently Implantable LDR CivaSheet®
Brief Title: Initial Feasibility Study to Treat Resectable Pancreatic Cancer With a Planar LDR Source
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CivaTech Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT005
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Pancreas Cancer; Cancer
Keywords: Whipple; brachytherapy; CivaSheet; CivaTech Oncology; radiation; intraoperative radiation; IORT; resectable pancreatic cancer; Pd-103
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Directional Brachytherapy Source Implant (Experimental): Patients undergoing a whipple procedure for pancreatic cancer will receive an implant at the time of surgery of the new CivaSheet directional brachytherapy device. The directional nature of the FDA cleared CivaSheet is expected to allow physicians to increase the radiation dose given to the surgical margin safely, reducing risk of recurrence without increasing radiation side effects.
  Interventions: Device: CivaSheet

INTERVENTIONS:
Device: CivaSheet — The FDA Cleared CivaSheet Directional Pd103 Brachytherapy Source is a planar radiation source which utilizes gold shielding in its construction. This device is radioactive on one side only, and is capable of safely delivering high doses of radiation to target areas even when placed directly adjacent to sensitive, healthy tissue or critical structures.

SUMMARY:
This is a Phase I evaluation to determine the usefulness of a new brachytherapy device that utilizes active components (Palladium-103) of standard devices in a novel configuration. This study may benefit resectable pancreatic cancer patients by reducing the radiation dose to adjacent critical structures, while giving a therapeutic dose to diseased tissue, such as at a surgical margin.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed informed consent
* Age >/= 18 years
* Biopsy confirmed adenocarcinoma pancreatic cancer
* Patient capable of undergoing anesthesia
* Patient is a surgical candidate
* Patient selected to undergo pancreatic cancer resection
* Patient will have known or suspected close/positive surgical margin
* Confirmed diagnosis of resectable pancreatic adenocarcinoma
* Will be prescribed standard Gemcitabine 1000 mg/m2 chemotherapy cycle

Exclusion Criteria:

* Pregnant or breast feeding
* Patient has metastatic disease
* Patient has had prior radiation therapy to the region for separate cancer
* Patient has had prior chemotherapy
* Any other invasive cancer in the past 5 years, except basal cell skin
* Recurrent or previously resected tumors
* Alcoholism/Drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Safety & Toxicity of Delivering Primary Radiation Therapy with CivaSheet using the CTCAE 4.0 scale | 1.5 years
  Patients with resectable pancreatic cancer who are undergoing pancreatic cancer resection will be monitored for safety & toxicities graded using the CTCAE 4.0 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- East Carolina University, Brody School of Medicine, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No